CLINICAL TRIAL: NCT02560974
Title: A Phase III Study Comparing Adjuvant Chemotherapy Consisting of Capecitabine/Oxaliplatin Versus Surgery Alone in Patients With Stage II (T1N2, T2N1, T3N0), IIIa (T2N2, T3N1, T4N0) and IIIb (T3N2) Gastric Adenocarcinoma
Brief Title: A Study of Capecitabine (Xeloda) in Combination Chemotherapy Versus Surgery Alone in Participants With Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO17527
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Capecitabine; Oxaliplatin

ARMS (2):
- Capecitabine + Oxaliplatin (Experimental): Patients will receive oral capecitabine (1000 mg/m^2 BID on Days 1 to 15 ) plus IV oxaliplatin (130 mg/m^2 on Day 1) during each 3-week cycle for up to 8 cycles (6 months).
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin
- Observation (No Intervention): Participants will not receive any treatment but will be seen regularly by a physician.

INTERVENTIONS:
Drug: Capecitabine — Capecitabine will be administered orally at 1000 mg/m^2 BID on Days 1 to 15 of a 3-week cycle, for 8 cycles.
  Other Names: Xeloda
  Arms: Capecitabine + Oxaliplatin
Drug: Oxaliplatin — Oxaliplatin will be administered as an IV infusion, 130 mg/m^2 on Day 1 of each 3-week cycle for 8 cycles.
  Arms: Capecitabine + Oxaliplatin

SUMMARY:
This study will compare capecitabine/oxaliplatin as adjuvant chemotherapy versus observation alone in chemotherapy-naive participants who have undergone potentially curative resection for gastric cancer. Participants will be randomized to either the chemotherapy arm or the observation arm. Capecitabine will be administered orally, 1000 milligrams per meter-squared (mg/m^2) twice daily (BID) on Days 1 to 15 of a 3-week cycle, for 8 cycles, and oxaliplatin will be administered as an intravenous (IV) infusion, 130 mg/m^2 every 3 weeks for 8 cycles. The anticipated time on study treatment in 6 months and the target sample size is 1024 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than or equal to (>=) 18 years of age
* Gastric adenocarcinoma, Stage II, IIIa or IIIb
* Potentially curative resection of tumor within 6 weeks prior to randomization
* Previously untreated with chemotherapy or radiotherapy

Exclusion Criteria:

* Serious concomitant medical illnesses that would limit life expectancy to less than (<) 5 years
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study
* Any evidence of metastatic disease (including presence of tumor cells in the ascites)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2006-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Disease-free survival rate | 3 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Incidence of adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (19):
- China (6):
  - Beijing
  - Fujian
  - Guangzhou
  - Shanghai
  - Shenyang
  - Tianjin
- South Korea (9):
  - Bundang City
  - Busan
  - Daegu
  - Gyeonggi-do
  - Incheon
  - Jeollabuk-do
  - Jeollanam-do
  - Seoul
  - Suwon
- Taiwan (4):
  - Changhua
  - Tainan
  - Taipei
  - Taoyuan District